CLINICAL TRIAL: NCT05416411
Title: Preoperative RESpiratory Training and MOBilization to Prevent Postoperative Pulmonary Complications in Patients Undergoing Thoracic Surgery (RESMOB): A Multi-center Randomized Controlled Trial
Brief Title: Preoperative RESpiratory Training and MOBilization to Prevent Postoperative Pulmonary Complications in Patients Undergoing Thoracic Surgery
Acronym: RESMOB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Emre Sertaç Bingül, Medical Doctor, Lecturer, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2018-2/39
Record Dates: First submitted 2022-06-08; First posted 2022-06-13 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Postoperative Complications; Procedure, Thoracic Surgical
Keywords: prehabilitation
MeSH Terms: conditions — Postoperative Complications | interventions — Walking

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Patients who are candidates for thoracic resection surgeries will be advised to stay active and quit smoking.
- Intervention group (Active Comparator): Patients who are candidates for thoracic resection surgeries will be handed a flow resistive device that helps inspiratory muscle training (2*30 repetitions a day for 7 days) and will be advised to walk 5000 steps a day.
  Interventions: Behavioral: Inspiratory muscle training

INTERVENTIONS:
Behavioral: Inspiratory muscle training — Patients will do inspiratory muscle training via a flow resistive device. Priorly, maximum inspiratory pressure will be measured. Afterwards, the training device will be set to 10% increased value of maximum inspiratory pressure (MIP), and the training will be completed two times and 30 repetitions a day during preoperative 7 days. Meanwhile patients will be advised to walk 5000 steps a day during the intervention period.
  Other Names: Walking (5000 steps/day)
  Arms: Intervention group

SUMMARY:
Postoperative pulmonary complications (PPCs) are the most frequent complications occurring in patients undergoing thoracic surgery and they are associated with prolonged hospital stay, decreased survival and expanding medical costs. Implementation of structured and supervised exercise programs including endurance training (ET), respiratory muscle training (RMT) or a combination of both, within the short waiting period before surgery, has been shown to enhance patients' physical fitness, to provide protective effects against PPCs and therefore to spare health care resources by shortening intensive care unit (ICU) and hospital lengths of stay. More recently, a simple intervention consisting in patient's instruction and education about modifiable risk factors, optimal breathing pattern and the impact of physical exercise has emerged as a simple alternative intervention prevent PPCs, although the evidence is inconclusive.

Therefore, the investigators propose a multicentre randomized, open, blinded end point controlled trial testing the hypothesis that preoperative education and instruction focused on breathing exercise and endurance training reduce the occurrence of PPCs in patients undergoing thoracic or abdominal surgery.

Patients with Intermediate-to-high risks factors for PPCs will be randomized on a 1:1 basis into an intervention arm and a usual care arm (Control group). In the Education group, patients will be asked to use a flow resistive device (One set of 30 repetitions, two times a day and to increase their daily physical activities (> 5'000 steps or equivalent) until surgery. Primary study endpoint will be the incidence of PPCs (e.g., atelectasis, pneumonia, respiratory failure) according to the European Perioperative Clinical Outcome definitions. Secondary outcomes will include non-respiratory complications, utilization of hospital resources (e.g., hospital length of stay, ICU admission),and preoperative changes in maximal inspiratory pressure [MIP]. Assuming a rate of 39% PPCs in the controls and a possible reduction to 26% in the intervention group, enrollment of 203 patients per group will provide 80% power with an alpha value of 0.05. Taking into account dropouts (5%) and in-hospital mortality rate (2%), a total of 436 surgical patients will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (> 18 years)
* Risk factors for PPCs (ARISCAT score >27)
* Elective intra-abdominal surgery or intrathoracic surgery via an open or minimally-invasive approach, expected to last > 120 min.

Exclusion Criteria:

* Patients unable to understand the instructions and/or to perform the proposed training program (i.e., poor comprehension, chest pain)
* COPD GOLD Grade III and IV, lung fibrosis, documented bullae, severe emphysema, pneumothorax
* Patient with chest pain or at risk of pneumothorax
* Previous lung surgery
* Bilateral lung procedures
* Emergent surgery or organ transplant
* Planned mechanical ventilation after surgery
* Uncontrolled asthma
* Coronary heart disease with angina grade 3 or 4 Canadian Cardiovascular Society
* documented pulmonary arterial hypertension >25mmHg mean pulmonary arterial pressure (PAP) at rest or > 40 mmHg systolic PAP (estimated by ultrasound)
* Documented or suspected neuromuscular disease (thymoma, myasthenia, myopathies, muscular dystrophies, others)
* Intracranial injury or tumor
* Persistent hemodynamnic instability, intractable shock
* Pregnancy (excluded by anamnesis and/or laboratory analysis)
* Enrollment in another interventional study or refusal of informed consent
* Presence of one of the adverse events, listed as PPCs (aspiration, respiratory failure, pneumonia, atelectasis, cardiopulmonary edema, pleural effusion, pneumothorax)
* Pleural surgery only, sympathectomy surgery only, chest wall surgery only, mediastinal surgery only, lung transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 436 (Estimated)
Dates: Start 2022-07-20 (Actual); Primary Completion 2024-07-10 (Estimated); Study Completion 2024-07-10 (Estimated)

PRIMARY OUTCOMES:
The incidence of postoperative pulmonary complications | Up to postoperative 5 days
  Postoperative pulmonary complications will be investigated during the postoperative 5 days. These complications are named according to the European Perioperative Clinical Outcome (EPCO) definitions (Respiratory failure, aspiration pneumonitis, pneumonia, ARDS, pneumothorax, atelectasis, bronchospasm)

SECONDARY OUTCOMES:
Preoperative MIP change | 7 days
  Maximum inspiratory pressure (MIP) will be measured during the enrollment and the training resistance will be set up according to this value. Once the training completed (after 7 days) another MIP measurement will be made
Length of stay in hospital | Up to 15 days
  Length of stay will be recorded as "days"
Visual Analog Scale thoracic rest pain | Up to 5 days
  Patients will be asked to describe their thoracic rest pain in a scale of 0 to 10
Visual Analog Scale thoracic coughing pain | Up to 5 days
  Patients will be asked to describe their thoracic coughing pain in a scale of 0 to 10
Visual Analog Scale dyspnea | Up to 5 days
  Patients will be asked to describe their dyspnea in a scale of 0 to 10

CONTACTS AND LOCATIONS:
Overall Officials: Emre S Bingul, MD, Principal Investigator — Istanbul University
Locations (3):
- Turkey (Türkiye) (3):
  - Acıbadem Mehmet Ali Aydınlar University, Faculty of Medicine, Istanbul
  - Istanbul University Istanbul Faculty of Medicine, Istanbul
  - Koc University, Faculty of Medicine, Istanbul

IPD SHARING:
Plan to Share IPD: Undecided